CLINICAL TRIAL: NCT03463785
Title: The Role of Race in the Pathogenesis of Obstructive Sleep Apnea: Asians Versus Caucasians
Brief Title: Does Race Make a Difference in Obstructive Sleep Apnea?
Status: Completed | Type: Observational
Sponsor: Academic Centre for Dentistry in Amsterdam (Other)
Collaborators: Shandong University (Other)
Responsible Party: Principal Investigator, Hui Chen, Dr., Academic Centre for Dentistry in Amsterdam
Other Study IDs: projectnummer 530-5CDP12
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: obstructive sleep apnea; race; upper airway; cone beam computed tomography
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chinese: Chinese mild or moderate OSA patients
  Interventions: Other: cone beam computed tomography
- Dutch: Dutch mild or moderate OSA patients
  Interventions: Other: cone beam computed tomography

INTERVENTIONS:
Other: cone beam computed tomography — The CBCT data sets of both the Chinese and Dutch OSA patients will be obtained using a NewTom 5G CBCT system (QR systems, Verona, Italy), according to the standard imaging protocol. The OSA patients will be treated with mandibular advancement device.
  Other Names: Mandibular advancement device (MAD)

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep-related breathing disorder, often associated with a compromised upper airway space and an increase in upper airway collapsibility. The anatomical and functional abnormalities of the upper airway play an important role in the pathogenesis of OSA. It is hypothesized that there is racial variation in the craniofacial characteristics among OSA patients. However, inter-race comparisons based on previous studies can be problematic due to variation in measurements, OSA definitions and the sample size. Besides, to our best knowledge, there is no studies that made direct inter-race comparisons in the upper airway anatomy. Therefore, studies on inter-race comparisons of the upper airway characteristics are needed to further understand the role of race in the upper airway anatomy of the OSA patients. This would provide more insights into the pathophysiology of OSA, and could result in the development of new effective treatment strategies for OSA patients.

DETAILED DESCRIPTION:
1. Patient recruitment In The Netherlands, the participants will be recruited from the sleep center of the Sint Lucas Andreas hospital in Amsterdam. The protocol of recruiting the patients from The Netherlands is approved by Medical Ethic Committee of AMC with the reference number NL44085.018.13/COSH.

   In China, the participants will be recruited from the sleep disorder center of dental school of Shandong University. The protocol of recruiting patients from China is approved by Medical Ethic Committee of Shandong University.

   Patients that fit the inclusion criteria will be approached to participate in the study in both The Netherlands and China.
2. Polysomnography (PSG) For the diagnosis of OSA, all the Chinese patients included in this study will undergo an overnight PSG recording (SOMNOscreenTM Plus PSG, Randersacker, Germany) at Qilu Hospital in Jinan, while all Dutch patients included in this study will undergo an overnight PSG recording (SOMNOscreenTM Plus PSG, Randersacker, Germany) in Amsterdam.

   PSG included the following variables: electroencephalogram, electro-oculogram, leg and chin electromyograms, electrocardiogram, pulse oximetry, body position, neck microphone, nasal cannula pressure transducer, and inductive plethysmography by means of thoracic and abdominal bands. The PSG recordings will be scored manually in a standard fashion. Apnea is defined as cession of airflow ≥90% for at least 10 seconds. Hypopnea is defined as a decrease in airflow of more than 30% for at least 10 seconds, and an oxygen desaturation greater than 4%. The mean apnea-hypopnea index (AHI) of the OSA group, defined as the number of apneas and hypopneas per hour of sleep.
3. Cone beam computed tomography (CBCT) In The Netherlands, CBCT scans of the OSA patients will be made at the department of Oral Radiology at ACTA. In China, CBCT scans of the OSA patients will be made at the department of Oral Radiology at Shandong University.

   The protocol for CBCT images in The Netherlands and China will be identical and is as follows: CBCT scans will be taken in the participants with the Frankfort plane perpendicular to the floor during their awake periods. The participants will be instructed not to swallow, speak, or do any motor response other than breathing during the CBCT procedure. The image detector and beam are positioned to maximize coverage of the upper airway from the level of nasal choanae to approximately the inferior edge of the fourth cervical vertebra.
4. Anatomical modeling of the upper airway Using Amira® (v4.1, Visage Imaging Inc., Carlsbad, CA, USA), the automatic process of the upper airway segmentation will be performed following the same protocol as in previous study. First, a voxel set is built to include all of the information of the upper airway; second, a new mask is built with its thresholds ranging from -1000 to -400; and third, the superior boundary (i.e., the plane across the PNS parallel to the FH plane) and the inferior boundary (i.e., the plane across the base of the epiglottis parallel to the FH plane) of the upper airway are selected in the corresponding axial planes and put into the voxel set. Finally, all of the slices between the upper and lower boundaries are selected and put into the voxel set.
5. Statistical analysis Whether the data are normally distributed was tested by the Shapiro-Wilk W Test. The Mann-Whitney-U test (for non-normally distributed variables) or Chi-squared test (for categorical variables) and the independent t-test (for normally distributed variables) are used to compare the differences in the demographic characteristics between the Chinese and Caucasian OSA patients. Patient characteristics that are significantly different between the two groups will be used as covariate(s) in the following between-group analysis. One-way multivariate analysis of covariance (MANCOVA) is used to compare the differences in anatomical and aerodynamic characteristics between the Chinese and Caucasian OSA patients. A significance level is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older;
2. Ability to speak, read, and write Dutch/Chinese;
3. Ability to follow-up;
4. Ability to use a computer with internet connection for online questionnaires;
5. Diagnosis with symptomatic mild or moderate OSA (5 ≤ apnea-hypopnea index (AHI) < 30);
6. Expected to maintain current lifestyle (sports, medicine, diet, etc.).

Exclusion Criteria:

1. Untreated periodontal problems, dental pain, and a lack of retention possibilities for a MAD;
2. Medication used/related to sleeping disorders;
3. Evidence of respiratory/sleep disorders other than OSA (eg. central sleep apnea syndrome);
4. Systemic disorders (based on medical history and examination; e.g. rheumatoid arthritis);
5. Temporomandibular disorders (based on the function examination of the masticatory system);
6. Medical history of known causes of tiredness by day, or severe sleep disruption (Insomnia, PLMS, Narcolepsy);
7. Known medical history of mental retardation, memory disorders, or psychiatric disorders.
8. Reversible morphological upper airway abnormalities (e.g. enlarged tonsils);
9. Inability to provide informed consent;
10. simultaneous use of other modalities to treat OSA;
11. Previous treatment with a MAD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the mild or moderate OSA patients with different racial background
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
the minimum cross-sectional area of the upper airway | within a week after taking CBCT scan of the patient
  measurement of the smallest area on the cross-sectional plane

SECONDARY OUTCOMES:
the anterior-posterior dimension of CSAmin | within a week after taking CBCT scan of the patient
  the longest distance of CSAmin anterior-posteriorly
the lateral dimension of CSAmin | within a week after taking CBCT scan of the patient
  the longest distance of CSAmin laterally
the volume of the upper airway | within a week after taking CBCT scan of the patient
  the volume of the upper airway (from hard palate to the base of epiglottis)
the length of the upper airway | within a week after taking CBCT scan of the patient
  the length of the upper airway (from hard palate to the base of epiglottis)

CONTACTS AND LOCATIONS:
Locations (2):
- Dentistry, Jinan, Shandong, China
- Dentistry, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the papers are accepted.
Access Criteria: The data will be shared with the researchers, who is interested in our project. The types of analyses used in the projected will be share via email to the corresponding authors.

REFERENCES:
- [Derived] Shi X, Chen H, Lobbezoo F, de Lange J, van der Stelt P, Berkhout E, Guo J, Ge S, Li G, Li Y, Aarab G. Comparison of the upper airway morphology between Dutch and Chinese adults with obstructive sleep apnea. Sleep Breath. 2023 Dec;27(6):2223-2230. doi: 10.1007/s11325-023-02834-z. Epub 2023 Apr 24. PMID 37093512